CLINICAL TRIAL: NCT05097664
Title: Ocular Manifestation and Related Risk Factors of Covid-19 Associated Mucormycosis: a Multicenter Study in Iran
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shiraz University of Medical Sciences (Other); Ahvaz Jundishapur University of Medical Sciences (Other); Iran University of Medical Sciences (Other); Mashhad University of Medical Sciences (Other); Tabriz University of Medical Sciences (Other); Guilan University of Medical Sciences (Other); Kermanshah University of Medical Sciences (Other); Shahid Beheshti University of Medical Sciences (Other); Semnan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohsen Pourazizi, Dr. Mohsen Pourazizi, Isfahan University of Medical Sciences
Other Study IDs: IR.MUI.MED.REC.1400.572
Record Dates: First submitted 2021-10-23; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Mucormycosis
Keywords: Coronavirus Disease-Associated Mucormycosis; COVID-19; Rhino-orbital-cerebral mucormycosis; Mucormycosis
MeSH Terms: conditions — COVID-19; Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) infection caused by the novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) may manifest as a variety of disease patterns, ranging from mild to life-threatening pneumonia.

Mucormycosis has been suspected to cause significant morbidity in infected people since the outbreak of the COVID-19 pandemic. Individuals who require hospitalization and intensive care are more vulnerable, as they have reached an advanced stage of their disease. Investigators will discuss the major risk factors, ocular presentation, and outcome of mucormycosis in individuals infected with SARS-CoV-2 in this study. From August 2021 to January 2022, a cross-sectional descriptive multicenter investigation would be conducted on patients with biopsy-confirmed mucormycosis and RTPCR confirmed COVID19. Demographic data, the time interval between COVID19 and mucormycosis, underlying systemic disorders, clinical characteristics, disease course, and outcomes would be analyzed.

DETAILED DESCRIPTION:
Investigators will achieved the following data from the participants:

1. Demographic
2. Past medical/habitual history
3. COVID-19 status and related risk factors
4. Mucormycosis status and related risk factors
5. Ocular examination and imaging
6. Follow-up

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of Mucormycosis in COVID-19 pandemic

Exclusion Criteria:

* People with acute or severely ill conditions that prevent them from ophthalmic examination.
* Patient, or legal representative opposing the pursuit of the research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Coronavirus Disease-Associated Mucormycosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-11-21 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Vision loss | 3 months
  Prevalence of Vision loss in COVID-19 patients with Mucormycosis co-infection

SECONDARY OUTCOMES:
Risk factors | 3 months
  Related risk factors for vision loss

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Pourazizi, M.D., Principal Investigator — Isfahan Eye Research Center
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

REFERENCES:
- [Derived] Eshraghi B, Khademi B, Bahmani Kashkouli M, Khataminia G, Kiarudi MY, Nabie R, Abounoori M, Chaibakhsh S, Ghahvehchian H, Rastegarnasab F, Parandin M, Zia Z, Karamirad S, Jafarpour S, Fakoor M, Varshochi M, Mirmohammadkhani M, Ramezani-Majd A, Janipour M, Mahdian Rad A, Shekarchian F, Manouchehri V, Sajjadi SMJ, Etezad Razavi M, Khosropour H, Forouhari A, Ebrahimi F, Pourazizi M. One-Year Patient Survival After COVID-19-Associated Rhino-Orbital-Cerebral Mucormycosis: A Multicenter Study. Mycopathologia. 2025 Jul 6;190(4):63. doi: 10.1007/s11046-025-00966-2. PMID 40619554